CLINICAL TRIAL: NCT06497179
Title: Impact of Handedness on Electromyographic Activity of Hand Muscles and Nerve Conduction Velocity During Mobile Phone Use in School-age Children
Brief Title: Effect of Handedness on Electromyographic Activity of Hand Muscles and Nerve Conduction Velocity During Use Mobil Phone in School Age Children
Status: Active, not recruiting | Type: Observational
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Rana Nabil Hussein Mohamed, lecturer of pediatric physical therapy in MTIU, MTI University
Other Study IDs: REC/211/MTI.PT/2406251
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Lateralization of the Brain Hemispheres

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Asymmetries in both physiology and anatomy at different levels of the central nervous system, which controls the upper extremities, are well-established. These asymmetries, related to handedness, are evident in the motor cortex and corticospinal tract. Moreover, variances have been identified in peripheral nervous pathways, including elevated sensory detection thresholds and increased conduction velocities in the motor nerve of the dominant arm.

Apart from disparities in the nervous system, differences also arise in the muscles. Prolonged preferential utilization of muscles on the dominant side of the body may lead to alterations in muscle fiber composition, characterized by a higher predominance of slow-twitch type I fibers.

Modern technology plays a key role in daily human life. This involves keeping pace with rapid changes in the field of communication technology. In this context, smartphones have become an essential part of life, not only in matters related to communication, but also as essential social accessories. As a result of this social involvement in communication technology, young children have become avid smartphones users. Holding a phone in hand needs support from fingers, flexion of hand and wrist, so holding the phone in same position for long periods can cause huge amount of stress on the structures present in the hand. This stress can cause injuries and damages in longer periods.

To address this objective, we will examine muscle synergies on the dominant sides in right-handed and left-handed participants while performing upper limb motor tasks. To accomplish this, we will conduct the following: Comparative analysis of motor and sensory nerve conduction velocities (radial, median, and ulnar) in right-handed and left-handed individuals during smartphone use. Comparison of hand muscle activation between right-handed and left-handed individuals during smartphone use.

DETAILED DESCRIPTION:
Handedness is a well-recognized behavioral phenomenon characterized by a preference for using one hand over the other. This study investigates the impact of handedness on electromyographic (EMG) activity of hand muscles and nerve conduction velocity during smartphone use.

This interventional parallel study included 70 participants (35 left-handed, 35 right-handed) aged 12 - 14 years inclusion criteria: normal BMI (16.5-24 kg/m²) no regular athletic activity, Participants shared the same socioeconomic level used the same smartphone model (6.7-inch touchscreen).

Exclusion criteria included:

peripheral nerve injury upper extremity movement limitations history of upper extremity fractures or deformities, neurological disorders such as peripheral neuropathy due to type I diabetes mellitus.

EMG activity and nerve conduction velocities (radial, median, and ulnar nerves) will be measured before and during smartphone use. Muscle activation will be assessed for the abductor pollicis longus (APL), extensor carpi radialis (ECR), flexor carpi ulnaris (FCU), and first dorsal interosseous muscles. Statistical analysis will be conducted to identify significant differences between left-handed and right-handed participants.

ELIGIBILITY:
Inclusion Criteria:

* normal BMI (16.5-24 kg/m²)
* no regular athletic activity, participated.
* Participants shared the same socioeconomic level
* used the same smartphone model (6.7-inch touchscreen)

Exclusion Criteria:

* peripheral nerve injury
* upper extremity movement limitations
* history of upper extremity fractures or deformities,
* neurological disorders such as peripheral neuropathy due to type I diabetes mellitus.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Seventy adolescents (35 left-handed, 35 right-handed) aged 12 to 14 years, with normal BMI (16.5-24 kg/m²) and no regular athletic activity, participated. Participants shared the same socioeconomic level and used the same smartphone model (6.7-inch touchscreen).
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Nerve Conduction Velocity | one day
  Nerves Assessed: Ulnar, median, and radial Phases: Phase 1: Pre-test without smartphone use. Phase 2: After 10 minutes of smartphone use. Consistency: Testing and laboratory environments will be kept constant. The same physiotherapist and neurophysiologist administered all tests. Measurements will be taken while participants used their dominant hand to operate the smartphone.
maximum voluntary isometric contraction (MVIC) | one day
  Muscle Activation Assessment for Flexor carpi ulnaris (FCU), extensor carpi radialis (ECR), abductor pollicis longus (APL), and first dorsal interosseous muscle. Positioning: Participants will sit on a chair with feet on the ground. Coupling gel will be applied to electrodes, straps will be used to prevent movement and wires will be kept loose. EMG machine functionality will be checked prior to use. MVIC measures and evaluates muscle strength and normalizes EMG data. Procedure: Explained to parents beforehand, with measurements will take on the same day. Peak force and target muscle force will be analyzed for MVIC. Data Analysis: Average Rectified EMG (ARV) will be used to measure muscle activity, as it is less variable compared to peak EMG variables. Changes in EMG signal indicating muscle fatigue included increased mean absolute value, amplitude, duration of muscle action potential, and a shift to lower frequencies.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of pysical therapy, MTI university, Cairo, Egypt